CLINICAL TRIAL: NCT00615927
Title: Phase II Study of Imatinib Mesylate Plus Hydroxyurea in the Treatment of Patients With Recurrent / Progressive Grade II Low-Grade Glioma
Brief Title: Phase II Imatinib + Hydroxyurea in Treatment of Patients With Recurrent/Progressive Grade II Low-Grade Glioma (LGG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008799
Record Dates: First submitted 2008-02-03; First posted 2008-02-14 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2012-12

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioblastoma; Gliosarcoma; glioblastoma multiforme (GBM); GBM; Imatinib Mesylate; Gleevec; Hydroxyurea; Droxia; Hydrea; Hydroxycarbamide; Imatinib; Brain tumor; Malignant brain tumor; Recurrent glioblastoma multiforme; Progressive glioblastoma multiforme
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Imatinib Mesylate; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Astrocytoma (Experimental): Grade II Astrocytoma
  Interventions: Drug: Imatinib Mesylate & Hydroxyurea
- Oligodendroglioma (Experimental): Grade II Oligodendroglioma or oligoastrocytomas
  Interventions: Drug: Imatinib Mesylate & Hydroxyurea

INTERVENTIONS:
Drug: Imatinib Mesylate & Hydroxyurea — Imatinib administered orally on daily. Imatinib is local irritant & must be taken in sitting position; mini of 2hrs should be allowed between last drug intake & going to bed. Imatinib doses 400mg/600mg administered once daily, whereas daily doses of 800mg/> administered as equally divided dose taken twice day. Dose for imatinib: Pts not receiving p450-inducing antiepileptic drugs: 400 mg/day. Pts receiving p450-inducing antiepileptic drugs: 500 mg twice day. It is recommended that pts take their prescribed imatinib mesylate at same time that they take their prescribed hydroxyurea, however, 30-60min interval between agents is acceptable if required for practical/other compliance issues.
  Hydroxyurea administered orally twice day. Dosing will begin on day 1 of cycle 1 & continue daily. Drug is approximately 80 percent bioavailable. Dose will be 500mg twice day for all pts.
  Other Names: Imatinib Mesylate-Gleevec; Hydroxyurea-Droxia-Hydrea-Hydroxycarbamide

SUMMARY:
Primary objective:

* To evaluate activity of imatinib mesylate and hydroxyurea among patients with progressive/recurrent grade II low-grade glioma (LGG) as measured by 12-month progression free survival

Secondary objectives:

* To evaluate progression-free survival (PFS), overall survival and objective response rate among patients with progressive/recurrent grade II LGG treated with imatinib mesylate plus hydroxyurea
* To assess safety and tolerability of imatinib mesylate + hydroxyurea in this population

DETAILED DESCRIPTION:
This is an open-label, single stage, uncontrolled, non-randomized Phase II study of continuous, daily doses of imatinib mesylate & hydroxyurea in adult patients with progressive/recurrent Grade II low-grade glioma (LGG). The treatment cycle is defined as imatinib mesylate & hydroxyurea administered daily for 28 days for purpose of scheduling evaluations. All patients who receive 1 or more doses of either imatinib mesylate or hydroxyurea will be evaluable for toxicity, whereas all patients who receive a minimum of 14 consecutive days of study regimen will be evaluable for response. Patients who discontinue therapy prior to receiving 14 consecutive days of study regimen will be regarded as ineligible for evaluation of response and will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade II LGG that is recurrent/progressive following prior surgical resection while on non-decreasing dose of corticosteroids
* > 25percent enlargement of bidimensional measure/new lesions on sequential imaging new &/or worsening neurologic deficits
* Patients with progressive/recurrent optic pathway tumors
* Patients have measurable disease on MRI/CT
* Interval of > 4 wks between prior external beam radiation therapy (XRT)/chemo,& enrollment on protocol unless there is unequivocal evidence of tumor progression & patient has recovered from all expected toxicities associated with prior therapy. Patients treated w chemo agents such as VP-16 who would normally be retreated after shorter intervals may be treated at usual starting time even if < 4 wks from last prior dose of chemo
* Patients not have had tumor biopsy < 1 wk/surgical resection < 2 wks prior to starting study drug
* Patients enrolling on arm B must be on > 1 enzyme inducing anticonvulsants for >2 wks prior to starting study drug
* Patients should be on non-increasing dose of steroids for > 7 days prior to obtaining baseline Gd-MRI of brain
* Patients should be on non-increasing dose of steroids for > 7 days prior to starting study drug
* Multifocal disease is eligible
* Age > 18 yrs old
* Karnofsky Performance Status (KPS) of > 60
* absolute neutrophil count (ANC) > 1.5 x 10 9/L
* Hgb > 9 g/dL
* Platelets > 100 x 10 9/L
* K ≥ lower limit of normal (LLN)/correctable with supplements
* Ca ≥ LLN/correctable with supplements
* P ≥ LLN/correctable with supplements
* aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) & Alanine transaminase (ALT)/ Serum Glutamic Pyruvate Transaminase (SGPT} < 2.5 x ULN
* Serum bilirubin < 1.5 x upper limit of normal (ULN)
* Serum creatinine < 1.5 x ULN/measured 24hr Creatinine Clearance > 50 mL/min/1.73m2
* Life expectancy ≥ 12wks
* Written informed consent obtained prior to screening procedures

Exclusion Criteria:

* Prior progressive disease/toxicity grade ≥ 3 with prior hydroxyurea therapy
* Prior treatment with imatinib/other platelet derived growth factor (PDGF)-directed therapy
* Excessive risk of bleeding as defined by stroke < 6 months, history of central nervous system (CNS)/intraocular bleed, or septic endocarditis
* Evidence of intratumor hemorrhage on pretreatment diagnostic imaging, except for stable post-operative gr1 hemorrhage
* Pregnant/breast feeding, /adults of reproductive potential not employing effective method of birth control
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in study
* Acute/chronic liver disease
* Confirmed diagnosis of HIV infection
* Impairment of GI function/GI disease that may significantly alter absorption of imatinib
* Patients taking Coumadin
* Patients have received investigational drugs < 2wks prior to entry on study/have not recovered from toxic effects of such therapy
* Patients have received biologic, immunotherapeutic/cytostatic agents < 1 wk prior to entry on study/have not recovered from toxic effects of such therapy
* Patient > 5 yrs free of another primary malignancy except: if other primary malignancy is not currently clinically significant/requiring active intervention, or if other primary malignancy is basal cell skin cancer/ cervical carcinoma in situ. Existence of any other malignant disease is not allowed
* Patients have had any surgery other than resection of brain tumor < 2 wks prior to entry on study/have not recovered from side effects of such therapy
* Patients unwilling to/unable to comply with protocol
* Active systemic bleeding, such as GI bleeding/gross hematuria
* Gr2 /> peripheral edema/central/systemic fluid collections
* Patients who enroll on arm A must have not received any EIAC for > 2 wks prior to starting study regimen
* Any of following exclusion criteria to MRI imaging:

  * Cardiac pacemaker
  * Ferromagnetic metal implants other than those approved as safe for use in magnetic resonance (MR) scanners
  * Claustrophobia
  * Obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Astrocytoma | Oligodendroglioma
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Astrocytoma | Oligodendroglioma | Total
Number analyzed (Participants) | 32 | 32 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 42.6 (16.6) | 46.6 (11.8) | 44.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: 12-month Progression Free Survival (PFS)
Description: Percentage of participants surviving twelve months from the start of cycle 1 without progression of disease. PFS was defined as the time from the cycle 1 start date to the date of the first documented progression according to modified Macdonald criteria, or to death due to any cause.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Astrocytoma | Oligodendroglioma
Number analyzed (Participants) | 32 | 32
percentage of participants | 43.8 [26.5 to 59.8] | 34.4 [18.8 to 50.6]

2. Secondary Outcome: Median Progression-free Survival
Description: Time in weeks from the start of cycle 1 to the date of first progression according to modified Macdonald criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: Time in weeks from the start of cycle 1 to the date of first progression according to modified Macdonald criteria or to death due to any cause, assessed up to 156 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Astrocytoma | Oligodendroglioma
Number analyzed (Participants) | 32 | 32
weeks | 43.5 [31.7 to 63.7] | 43.3 [24.9 to 53.6]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Time in weeks from the start of cycle 1 to date of death due to any cause. Patients alive at last follow-up are censored as of that follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: Time in weeks from the start of cycle 1 to date of death due to any cause, assessed up to 156 weeks
Population: Median overall survival was not estimable for either arm as not enough events of death occurred
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Astrocytoma | Oligodendroglioma
Number analyzed (Participants) | 32 | 32
weeks | NA [NA to NA] — Median overall survival was not estimable for either arm as not enough events of death occurred. | NA [NA to NA] — Median overall survival was not estimable for either arm as not enough events of death occurred.

4. Secondary Outcome: Objective Response Rate
Description: Number of participants with an objective response (complete response or partial response) based on modified Macdonald criteria.
Time Frame: 156 weeks
Measure: Number; unit: participants
Arm/Group | Astrocytoma | Oligodendroglioma
Number analyzed (Participants) | 32 | 32
participants | 0 | 0

5. Secondary Outcome: Safety and Tolerability of Gleevec + Hydroxyurea in Patients With Low-grade Gliomas
Description: The number of patients experiencing any serious adverse event or other (non-serious) adverse event during the study participation.
Time Frame: 156 weeks
Measure: Number; unit: participants
Arm/Group | Astrocytoma | Oligodendroglioma
Number analyzed (Participants) | 32 | 32
participants
  Experienced any Serious Adverse Event | 10 | 3
  Experienced any (non-serious) Adverse Event | 28 | 28

ADVERSE EVENTS:
Time Frame: 156 weeks
Description: All adverse events were gathered for the study using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, but were converted to CTCAE version 4.0 for entry into ClinicalTrials.gov.
Arm/Group | Astrocytoma | Oligodendroglioma
Serious Adverse Events (participants affected / at risk) | 10/32 | 3/32
Other Adverse Events (participants affected / at risk) | 28/32 | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Astrocytoma (N=32) | Oligodendroglioma (N=32)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Cardiac disorders-Other, specify: Coronary artery disease (Cardiac disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Death NOS (General disorders) | 2 | 0
Edema face (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Psychosis (Psychiatric disorders) | 0 | 1
Renal and urinary disorders-Other, specify: Renal and splenic infarcts (Renal and urinary disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Astrocytoma (N=32) | Oligodendroglioma (N=32)
Anemia (Blood and lymphatic system disorders) | 3 | 2
Blurred vision (Eye disorders) | 10 | 8
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 6 | 7
Mucositis oral (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 10 | 7
Vomiting (Gastrointestinal disorders) | 2 | 1
Edema limbs (General disorders) | 3 | 0
Fatigue (General disorders) | 16 | 15
Fever (General disorders) | 0 | 2
Pain (General disorders) | 3 | 2
Bronchial infection (Infections and infestations) | 0 | 2
Infections and infestations-Other, specify: Head cold (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 3 | 0
Skin infection (Infections and infestations) | 2 | 0
Upper respiratory infection (Infections and infestations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 3 | 7
Platelet count decreased (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Ataxia (Nervous system disorders) | 9 | 8
Cognitive disturbance (Nervous system disorders) | 4 | 9
Depressed level of consciousness (Nervous system disorders) | 3 | 6
Dizziness (Nervous system disorders) | 6 | 6
Dysphasia (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 10 | 16
Memory impairment (Nervous system disorders) | 5 | 6
Nervous system disorders-Other, specify: Mood Alteration, NOS (Nervous system disorders) | 1 | 3
Peripheral motor neuropathy (Nervous system disorders) | 8 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 7
Seizure (Nervous system disorders) | 7 | 8
Tremor (Nervous system disorders) | 4 | 2
Agitation (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 2
Confusion (Psychiatric disorders) | 6 | 5
Depression (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 6 | 7
Libido decreased (Psychiatric disorders) | 0 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 2
Reproductive system and breast disorders-Other, specify: Sexual Dysfunction (Reproductive system and breast disorders) | 4 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No